CLINICAL TRIAL: NCT02462798
Title: Does Sourdough Fermentation Improve Iron Uptake From Whole Grain Rye Bread?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Chalmers0002
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Iron Bioavailability; Anaemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole grain rye bread (Placebo Comparator): Whole grain rye bread, 200 g/d. Control intervention.
  Interventions: Other: Whole grain rye bread
- Whole grain sourdough rye bread (Experimental): Whole grain rye bread, 200 g/d. Experimental intervention.
  Interventions: Other: Whole grain sourdough rye bread

INTERVENTIONS:
Other: Whole grain rye bread — Whole grain rye bread baked without sourdough fermentation (normal yeast-based fermentation)
  Arms: Whole grain rye bread
Other: Whole grain sourdough rye bread — Whole grain rye bread fermented with sourdough culture before baking
  Arms: Whole grain sourdough rye bread

SUMMARY:
Iron deficiency anaemia is a major problem for women worldwide. Cereal foods are a major source of iron, but much of this is not bioavailability due to it being bound by the high amounts of phytate present in cereals. Destruction of phytate by the phytase enzyme can release iron and increase its bioavailability. In a human cell model of iron uptake, sourdough fermentation, which included activation of phytase, the enzyme that breaks down phyate, led to improved iron bioavailability. This clinical trial will attempt to demonstrate that this concept also works in humans

ELIGIBILITY:
Inclusion Criteria:

* Healthy women under 50 years old

Exclusion Criteria:

* Pregnancy or breast feeding
* Use of mineral or other dietary supplements
* Use of medical or recreational drugs
* Donation of blood within the previous 3 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Serum ferritin | 12 week values corrected for baseline
Serum transferrin receptor | 12 week values corrected for baseline
Haemoglobin | 12 week values corrected for baseline